CLINICAL TRIAL: NCT04000438
Title: Randomized, Placebo-Controlled, Proof of Concept Study to Evaluate the Efficacy on Cervical Ripening, Safety, Tolerability and Dose Response of SC Administered Tafoxiparin in Term Pregnant, Nulliparous Women With an Unripe Cervix Undergoing Labor Induction
Brief Title: Effect of Tafoxiparin on Cervical Ripening and Induction of Labor in Term Pregnant Women With an Unripe Cervix
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dilafor AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PPL17; 2019-000620-17 (EudraCT Number)
Record Dates: First submitted 2019-06-14; First posted 2019-06-27 (Actual); Results first posted 2025-04-09 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-03

CONDITIONS: Labor Onset and Length Abnormalities
Keywords: Priming of labor; Unripe cervix; Home treatment; Cervical ripening; Labor induction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental DF01 high dose (Experimental): The subject receives sc injections once daily for up to 7 days until labor induction or spontaneous onset of labor.
  Interventions: Drug: DF01
- Experimental: DF01 medium dose (Experimental): The subject receives sc injections once daily for up to 7 days until labor induction or spontaneous onset of labor.
  Interventions: Drug: DF01
- Experimental: DF01 low dose (Experimental): The subject receives sc injections once daily for up to 7 days until labor induction or spontaneous onset of labor.
  Interventions: Drug: DF01
- Placebo comparator: PL1 (Placebo Comparator): The subject receives sc injections once daily for up to 7 days until labor induction or spontaneous onset of labor.
  Interventions: Drug: PL1

INTERVENTIONS:
Drug: DF01 — DF01: The subject receives sc injections of tafoxiparin solution once daily for up to 7 days until spontaneous onset of labor or ripe cervix (Amniotomy/oxytocin without restriction).If not enough ripening cervical ripening according to clinical practice with intracervical ballon/prostaglandins
  Other Names: tafoxiparin
  Arms: Experimental DF01 high dose; Experimental: DF01 low dose; Experimental: DF01 medium dose
Drug: PL1 — DF01: The subject receives sc injections of placebo solution once daily for up to 7 days until spontaneous onset of labor or ripe cervix (Amniotomy/oxytocin without restriction).If not enough ripening cervical ripening according to clinical practice with intracervical ballon/prostaglandins
  Other Names: Placebo
  Arms: Placebo comparator: PL1

SUMMARY:
The study is designed as a randomized, Double-Blind, Placebo-Controlled, Parallel-Group Proof of Concept Study (section A) with a conditional dose finding follow up (Section B) to Evaluate the Efficacy on Cervical ripening, Safety, Tolerability and dose response of Subcutaneously Administered Tafoxiparin in Term Pregnant, Nulliparous Women with an unripe cervix undergoing Labor Induction. If the efficacy and safety profiles of Section A are conclusive in favor of tafoxiparin, the study will continue by adding two additional tafoxiparin dose groups in Section B.

DETAILED DESCRIPTION:
Primary objective:

To assess the efficacy of tafoxiparin on cervical ripening.

Secondary objective:

To assess the maternal and neonatal safety, tolerability and dose response of tafoxiparin as a supplement therapy in term pregnant, nulliparous women with an unripe cervix undergoing labor induction

Methodology:

Term pregnant, nulliparous women with unripe cervix and planned for labor induction are potential study patients unless enrolled in another study. Subjects may be preinformed about the study through the use of advertisement or information at the physician/midwife visits during pregnancy and at the hospital admission.

The whole study includes the following steps:

Screening and Baseline including informed consent and randomization Study treatment and Induction of Labor Labor Discharge

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women of ≥18 and ≤ 64 years of age
* Nulliparous
* Unripe cervix with ≤ 4points according to Bishop/Westin score (0-10 points scale)
* Planned for labor induction after 4-7 days of IMP treatment
* Examples of diagnosis as a basis for induction:

  * Post term pregnancy (40-41 weeks of gestation)
  * Gestational diabetes
  * Diabetes type 1 - well controlled
  * Pre-eclampsia (BP diastolic <100, systolic <140)
  * Hypertension - well controlled
  * Hepatosis (without clinically significantly elevated serum bile acids)
  * Maternal age ≥ 40 years
  * Humanitarian-psycho social reasons
  * Oligohydramnios
* Gestational age > 37 weeks confirmed by ultrasound before 21 weeks of gestation
* Singleton pregnancy
* Subject is, as per the discretion of the Investigator, able to comply with the requirements of the protocol including an ability to be present at all required controls
* Subject can understand and sign an informed form
* Provision of written informed consent

Exclusion Criteria:

* Subjects who are unable to understand the written and verbal instructions in local language
* Breech presentation and other abnormal fetal presentations
* Previous uterine scar
* Spontaneous rupture of membranes at inclusion
* Pathologic CTG at inclusion
* Fetal estimated weight > 2SD of normal fetal estimated weight earlier diagnosed by ultrasound and documented in patient record
* Mother's BMI > 35 at early pregnancy
* Known IUGR defined as ≤ 2SD of normal
* Presence of eclampsia
* Severe Pre-eclampsia
* HELLP syndrome (hemolysis, elevated liver enzymes, and low platelets)
* Clinically significant vaginal bleeding in need of hospitalization in the third trimester
* Placenta previa
* Previously known coagulation disorders (Leiden, heterozygote - OK)
* Current use of any drugs that interfere with hemostasis (including heparin /LMWH, direct oral anti-coagulant medication, non-steroidal anti-inflammatory drugs (NSAID) compounds and vitamin K antagonists.)
* Current use of acetylsalicylic acid (ASA) compounds or use within the week preceding inclusion
* Diagnosed with HIV or Acute hepatitis
* Known history of allergy to standard heparin and/or LMWH heparin
* History of heparin-induced thrombocytopenia
* Current drug or alcohol abuse which in the opinion of the Investigator should preclude participation in the study.
* Current participation in other interventional medicinal treatment studies
* Subject has a fear of needles which is believed by the Investigator to affect study medication compliance

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 365 (Actual)
Dates: Start 2019-06-21 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gunvor Ekman-Ordeberg, MD, PhD, Study Chair, CMO, Study Chair — CMO
Locations (7):
- Finland (2):
  - Naistenklinikka (HUS), Helsinki
  - Tampere University Hospital, Tampere
- Sweden (5):
  - Kvinnokliniken Universitetssjukhuset Linköping, Linköping
  - Lund University Hospital, Lund
  - Kvinnokliniken Skaraborgs Sjukhus, Skövde
  - Kvinnokliniken Södersjukhuset, Stockholm
  - Förlossningsavdelningen Akademiska Universitetssjukhuset, Uppsala

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Number of subjects screened/enrolled: 365 Number of subjects started: 348
  Reason: 17 subjects did not pass inclusion/exclusion
Groups:
- Experimental DF01 High Dose; Experimental: DF01 Medium Dose; Experimental: DF01 Low Dose: The subject receives sc injections once daily for up to 7 days until labor induction or spontaneous onset of labor.
  DF01: The subject receives sc injections of tafoxiparin solution once daily for up to 7 days until spontaneous onset of labor or ripe cervix (Amniotomy/oxytocin without restriction).If not enough ripening cervical ripening according to clinical practice with intracervical ballon/prostaglandins
- Placebo Comparator: PL1: The subject receives sc injections once daily for up to 7 days until labor induction or spontaneous onset of labor.
  PL1: The subject receives sc injections of placebo solution once daily for up to 7 days until spontaneous onset of labor or ripe cervix (Amniotomy/oxytocin without restriction).If not enough ripening cervical ripening according to clinical practice with intracervical ballon/prostaglandins
Period: Overall Study
Arm/Group | Experimental DF01 High Dose | Experimental: DF01 Medium Dose | Experimental: DF01 Low Dose | Placebo Comparator: PL1
Started | 91 | 85 | 83 | 89
Completed | 90 | 85 | 82 | 86
Not Completed | 1 | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental DF01 High Dose | Experimental: DF01 Medium Dose | Experimental: DF01 Low Dose | Placebo Comparator: PL1 | Total
Number analyzed (Participants) | 91 | 85 | 83 | 89 | 348
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 91 | 85 | 83 | 89 | 348
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.2 (4.34) | 31.4 (4.22) | 31.6 (5.28) | 31.3 (5.04) | 31.4 (4.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 85 | 83 | 89 | 348
  Male | 0 | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 27 | 30 | 26 | 28 | 111
  Finland | 64 | 55 | 57 | 61 | 237

OUTCOME MEASURES:

1. Primary Outcome: Cervical Ripening Rate, Measured by Bishop Score - Slope
Description: Cervical ripening rate during up to the first seven days of treatment, measured by Bishop Score - Slope.
  Bishop score is an Assessment of the cervical stage by its: dilatation, position, effacement and consistency.
  The score was calculated as the sum of the following 5 categories where each category is scored between 0-2:
  * Fetal station (0-2)
  * Cervical diameter at inner meatus (0-2)
  * Cervical effacement (0-2)
  * Consistency at inner meatus (0-2)
  * Cervical position (0-2) Graded from 0-10, Bishop score of ≤ 4 is unripe and ≥ 6 is ripe.
  Bishop score was measured daily from start of treatment up until 7 days. The cervical ripening rate was calculated from the slope of the curve (score/day) when plotting Bishop score against days of treatment.
Time Frame: Daily measures of Bishop Score from start of study drug administration until delivery (up to 7 days).
Measure: Mean (Standard Deviation); unit: Slope (Bishop Score/day)
Groups:
- Experimental DF01 High Dose: The subject receives sc injections once daily for up to 7 days until labor induction or spontaneous onset of labor.
  DF01: TThe subject receives sc injections of tafoxiparin solution once daily for up to 7 days until spontaneous onset of labor or ripe cervix (Amniotomy/oxytocin without restriction).If not enough ripening cervical ripening according to clinical practice with intracervical ballon/prostaglandins.
Arm/Group | Experimental DF01 High Dose | Experimental: DF01 Medium Dose | Experimental: DF01 Low Dose | Placebo Comparator: PL1
Number analyzed (Participants) | 91 | 85 | 83 | 88
Slope (Bishop Score/day) | 0.86 (0.062) | 0.81 (0.062) | 0.78 (0.061) | 0.62 (0.060)

ADVERSE EVENTS:
Time Frame: From first dose to until discharge from hospital, an average of 9.3 days.
Groups:
- Placebo Comparator: PL1: The subject receives sc injections once daily for up to 7 days until labor induction or spontaneous onset of labor.
  DF01: The subject receives sc injections of placebo solution once daily for up to 7 days until spontaneous onset of labor or ripe cervix (Amniotomy/oxytocin without restriction).If not enough ripening cervical ripening according to clinical practice with intracervical ballon/prostaglandins
Arm/Group | Experimental DF01 High Dose | Experimental: DF01 Medium Dose | Experimental: DF01 Low Dose | Placebo Comparator: PL1
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/85 | 0/83 | 0/88
Serious Adverse Events (participants affected / at risk) | 6/91 | 7/85 | 2/83 | 2/88
Other Adverse Events (participants affected / at risk) | 52/91 | 54/85 | 54/83 | 47/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental DF01 High Dose (N=91) | Experimental: DF01 Medium Dose (N=85) | Experimental: DF01 Low Dose (N=83) | Placebo Comparator: PL1 (N=88)
Amniotic cavity infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postpartum sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bradycardia foetal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Total bile acids increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental DF01 High Dose (N=91) | Experimental: DF01 Medium Dose (N=85) | Experimental: DF01 Low Dose (N=83) | Placebo Comparator: PL1 (N=88)
Perineal injury (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 17 (17) | 21 (21) | 4 (4)
Bradycardia foetal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 6 (6) | 1 (3) | 0 (0)
Tachycardia foetal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Uterine atony (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Retained placenta or membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Labour pain (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Inferior vena cava syndrome (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Symphysiolysis (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Foetal hypokinesia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Transient tachypnoea of the newborn (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prolonged labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Placental calcification (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic haematoma obstetric (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine hyperstimulation (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine contractions abnormal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 8 (8) | 9 (9) | 11 (11) | 7 (7)
Injection site pain (General disorders) | 8 (14) | 2 (2) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 4 (4) | 5 (6) | 0 (0)
Injection site bruising (General disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Injection site discolouration (General disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Injection site swelling (General disorders) | 2 (3) | 2 (2) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (2)
Injection site erythema (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injection site pruritus (General disorders) | 1 (5) | 1 (1) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Malaise (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site warmth (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Puncture site haemorrhage (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 6 (7) | 2 (2) | 6 (6)
Vomiting (Gastrointestinal disorders) | 2 (2) | 6 (6) | 5 (5) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3) | 4 (4)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 6 (6) | 7 (7) | 8 (10) | 5 (5)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Insomnia (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Post lumbar puncture syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aura (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 6 (6) | 10 (10) | 6 (6) | 7 (8)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glycosuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukocyturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 6 (6) | 2 (3) | 4 (4) | 3 (3)
Hepatic enzyme increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Foetal monitoring abnormal (Investigations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Blood lactic acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood lactate dehydrogenase abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual analogue scale (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal injury (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 1 (1) | 5 (5)
Cervical discharge (Reproductive system and breast disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vaginal haematoma (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amniotic cavity infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Genital herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 6 (6) | 3 (3) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Thymus enlargement (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Haemorrhage (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Epistaxis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulval haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder catheterisation (Surgical and medical procedures) | 6 (6) | 0 (0) | 0 (0) | 3 (3)
Caesarean section (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Episiotomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epidural anaesthesia (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Skin discolouration (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal sphincter injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaesthetic complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obstetric procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abnormal sensation in eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-15): https://cdn.clinicaltrials.gov/large-docs/38/NCT04000438/Prot_SAP_000.pdf